CLINICAL TRIAL: NCT04091048
Title: Optimize PRO Transcatheter Aortic Valve Replacement Post Market Study
Brief Title: Optimize PRO Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18051EVR008
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Aortic Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Primary Cohort
  Interventions: Device: Evolut™ PRO and Evolut™ PRO+ System (Evolut™ FX System for the addendum)

INTERVENTIONS:
Device: Evolut™ PRO and Evolut™ PRO+ System (Evolut™ FX System for the addendum) — Aortic valve replacement

SUMMARY:
The purpose of this study is to collect clinical evidence on valve performance and procedural outcomes associated with an "optimized" TAVR care pathway and post-TAVR conduction disturbance pathway while using the Evolut™ PRO and Evolut™ PRO+ devices.

The purpose of the addendum is to collect post-market clinical evidence on valve performance and procedural outcomes associated with the Evolut FX Device.

DETAILED DESCRIPTION:
This is a post market, multi-center (sites in US/CAN/EMEA/ANZ), prospective, non-randomized study.

The addendum is a post market, multi-center (sites in US only), prospective, non-randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable candidate for treatment with the Evolut™ PRO or Evolut™ PRO+ system (FX system for the addendum where applicable) in accordance with the Instructions for Use and local regulations;
* Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater;
* Subject and the treating physician agree that the subject will return for all required post procedure follow-up visits;
* Anatomically suitable for transfemoral TAVR with the Medtronic TAVR system;
* Subject meets the legal minimum age to provide Informed Consent based on local regulatory requirements.

Exclusion Criteria:

* Contraindicated for treatment with the Evolut™ PRO or Evolut™ PRO+ or FX system (where applicable) in accordance with the Instructions for Use
* Anatomically not suitable for the Evolut™ PRO or Evolut™ PRO+ or FX system (where applicable);
* Previous aortic valve replacement
* Reduced ventricular function with left ventricular ejection fraction (LVEF) <35% as measured by resting echocardiogram;
* Frailty assessments identify:

  * Subject is <80 years of age and three or more of the following apply; OR subject is > 80 years of age and two or more of the following apply

    * Wheelchair bound
    * Resides in an institutional care facility (e.g. nursing home, skilled care center)
    * Body Mass Index <20kg/m2
    * Grip strength <16kg
    * Katz Index score ≤4
    * Albumin <3.5 g/dL
* Bicuspid valve verified;
* Aortic root angulation (angle between plane of aortic valve annulus and horizontal plane/vertebrae) > 70°.
* Implanted with pacemaker or ICD;
* Prohibitive left ventricular outflow tract calcification;
* Estimated life expectancy of less than 12 months due to associated non- cardiac co-morbid conditions;
* Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent, adherence to the protocol required follow-up exams;
* Currently participating in an investigational drug or another device trial (excluding registries);
* Need for emergency surgery for any reason.
* Subject is less than legal age of consent, legally incompetent, or otherwise vulnerable*.

  * Notes: Vulnerable subjects include individuals whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate. EXAMPLE Individuals with lack of or loss of autonomy due to immaturity or through mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, and those incapable of giving informed consent. Other vulnerable subjects include, for example, members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces, and persons kept in detention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients with symptomatic native aortic valve stenosis that necessitates valve replacement who meet the criteria for on-label use of the Evolut™ PRO or Evolut™ PRO+ (and FX system for the addendum where applicable) system in accordance with Instructions for Use and local regulations.
Sampling Method: Non-Probability Sample
Enrollment: 1127 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Yakubov, MD, Principal Investigator — OhioHealth; Kendra Grubb, MD, Principal Investigator — Emory University; Josep Rodés-Cabau, MD, Study Chair — Laval University; Suneet Mittal, MD, Study Chair — Valley Health System; Tamim Nazif, MD, Study Chair — Columbia - New York Presbyterian; Hemal Gada, MD, Study Chair — UPMC Pinnacle; Douglas Fraser, MD, Study Chair — Manchester Royal Infirmary
Locations (60):
- United States (37):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - California Pacific Medical Center - Sutter Health, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - St. Vincent's Hospital / Cardiology Associates of Fairfield County, P.C., Norwalk, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - St. John's Hospital/Prarie Education and Research Cooperative, Springfield, Illinois
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Abbott Northwestern Hospital (Minneapolis Heart), Minneapolis, Minnesota
  - Providence St. Patrick Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - The Mount Sinai Hospital, New York, New York
  - New York Presbyterian - Columbia University Medical Center, New York, New York
  - Vassar Brother's Medical Center, Poughkeepsie, New York
  - St. Francis Hospital, Roslyn, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Ohio Health Research Institute, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - The Heart Hospital - Baylor Plano, Plano, Texas
  - Dixie Regional Medical Center Intermountain, St. George, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Charleston Medical Center, Charleston, West Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Australia (7):
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside West
  - Monash Hospital, Clayton
  - Austin Hospital, Heidelberg
  - Fiona Stanley Hospital, Murdoch
  - John Hunter Hospital, Newcastle
  - Saint Vincents Hospital Sydney, Sydney
- Belgium (2):
  - ZNA Middelheim, Antwerp
  - St Jan Hospital, Bruges
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Laval University Institute of Cardiology and Respirology of Quebec, Québec, Quebec
- France (2):
  - Hôpitaux Universitaires - Hôpital Henri Mondor, Créteil
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac
- Universitätsklinikum Ulm, Ulm, Germany
- Ireland (2):
  - Mater Private Hospital, Dublin
  - Galway University Hospitals - University Hospital Galway (UHG), Galway
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (2):
  - Fondazione Poliambulanza, Brescia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Hospital Universitario Central de Asturas, Oviedo, Spain
- Akademiska Sjukhuset, Uppsala, Sweden
- United Kingdom (2):
  - Royal Victoria Hospital - Belfast Health and Social Care Trust, Belfast
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grubb KJ, Gada H, Mittal S, Nazif T, Rodes-Cabau J, Fraser DGW, Lin L, Rovin JD, Khalil R, Sultan I, Gardner B, Lorenz D, Chetcuti SJ, Patel NC, Harvey JE, Mahoney P, Schwartz B, Jafar Z, Wang J, Potluri S, Vora AN, Sanchez C, Corrigan A, Li S, Yakubov SJ. Clinical Impact of Standardized TAVR Technique and Care Pathway: Insights From the Optimize PRO Study. JACC Cardiovasc Interv. 2023 Mar 13;16(5):558-570. doi: 10.1016/j.jcin.2023.01.016. PMID 36922042

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Protocol: Evolut™ PRO and Evolut™ PRO+ System: Aortic valve replacement
- FX Addendum: Evolut™ FX System: Aortic valve replacement
Period: Overall Study
Arm/Group | Main Protocol | FX Addendum
Started | 928 | 199
Completed | 653 | 151
Not Completed | 275 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Protocol | FX Addendum | Total
Number analyzed (Participants) | 653 | 151 | 804
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Results of the Main Protocol and FX Addendum are analyzed separately.
  years
    Main Protocol: number analyzed (Participants) | 653 | 0 | 653
    Main Protocol | 79.1 (6.5) |  | 79.1 (6.5)
    FX Addendum Cohort: number analyzed (Participants) | 0 | 151 | 151
    FX Addendum Cohort |  | 78.3 (7.1) | 78.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Results of the Main Protocol and FX Addendum are analyzed separately.
  Participants
    Main Protocol: number analyzed (Participants) | 653 | 0 | 653
    Main Protocol: Female | 307 |  | 307
    Main Protocol: Male | 346 |  | 346
    FX Addendum: number analyzed (Participants) | 0 | 151 | 151
    FX Addendum: Female |  | 67 | 67
    FX Addendum: Male |  | 84 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Main Protocol: Ethnicity and race are reported only by United States, Canada, Australia and New Zealand (n=451). Not reported for Europe, Middle East, and Africa (EMEA [n=202]).
  Results of the Main Protocol and FX Addendum are analyzed separately.
  Participants
    Main Protocol: number analyzed (Participants) | 451 | 0 | 451
    Main Protocol: American Indian or Alaska Native | 1 |  | 1
    Main Protocol: Asian | 1 |  | 1
    Main Protocol: Black or African American | 11 |  | 11
    Main Protocol: Native Hawaiian or Other Pacific Islander | 1 |  | 1
    Main Protocol: White | 432 |  | 432
    Main Protocol: Other | 5 |  | 5
    FX Addendum: number analyzed (Participants) | 0 | 151 | 151
    FX Addendum: American Indian or Alaska Native |  | 1 | 1
    FX Addendum: Asian |  | 0 | 0
    FX Addendum: Black or African American |  | 6 | 6
    FX Addendum: Native Hawaiian or Other Pacific Islander |  | 2 | 2
    FX Addendum: White |  | 141 | 141
    FX Addendum: Other |  | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Results of the Main Protocol and FX Addendum are analyzed separately
  kg/m^2
    Main Protocol: number analyzed (Participants) | 653 | 0 | 653
    Main Protocol | 29.6 (5.9) |  | 29.6 (5.9)
    FX Addendum: number analyzed (Participants) | 0 | 151 | 151
    FX Addendum |  | 30.2 (6.0) | 30.2 (6.0)
NYHA [Count of Participants; unit: Participants] — New York Heart Association (NYHA):
  Class I:No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue palpitation, shortness or breath or chest pain.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  Class IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort. Population: Results of the Main Protocol and FX Addendum are analyzed separately.
  Participants
    Main Protocol: number analyzed (Participants) | 653 | 0 | 653
    Main Protocol: NYHA I | 0 |  | 0
    Main Protocol: NYHA II | 374 |  | 374
    Main Protocol: NYHA III | 256 |  | 256
    Main Protocol: NYHA IV | 23 |  | 23
    FX Addendum: number analyzed (Participants) | 0 | 151 | 151
    FX Addendum: NYHA I |  | 1 | 1
    FX Addendum: NYHA II |  | 110 | 110
    FX Addendum: NYHA III |  | 38 | 38
    FX Addendum: NYHA IV |  | 2 | 2
STS Score [Mean (Standard Deviation); unit: Mean] — The Society of Thoracic Surgeons (STS) Score is a score that represents the risk of operative mortality, major morbidity, and complications for adult cardiac surgeries.
  A total STS Score, presented as a risk probability on a scale of 0-100%, is calculated based on patient characteristics.
  The STS Score is calculated before a patient undergoes the transcatheter aortic valve replacement (TAVR) index procedure in the study, and a higher STS Score means a patient is at higher risk for surgery. Population: Results of the Main Protocol and FX Addendum are analyzed separately.
  Mean
    Main Protocol: number analyzed (Participants) | 653 | 0 | 653
    Main Protocol | 3.2 (2.5) |  | 3.3 (2.3)
    FX Addendum: number analyzed (Participants) | 0 | 151 | 151
    FX Addendum |  | 3.1 (2.0) | 3.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality or All-stroke
Description: All-cause mortality or all-stroke at 30 days.
Time Frame: 30 days post procedure
Population: The attempted implant set was the basis for the primary outcome measure for the Main Protocol and FX Addendum.
  The attempted implant set consists of all enrolled subjects with an attempted TAVR implant procedure, defined as when the subject is brought into the procedure room and any of the following have occurred: anesthesia or conscious sedation administered, vascular line placed, TEE placed, or any monitoring line placed.
  Main Protocol and FX Addendum results are analyzed separately.
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Main Protocol | FX Addendum
Number analyzed (Participants) | 653 | 151
Percent of Participants (K-M Rate) | 5.1 | 2.7

2. Secondary Outcome: Length of Stay
Description: Median days from index procedure to discharge
Time Frame: Through discharge up to 7 days post index procedure.
Population: The basis for the length of stay secondary outcome measure was the per-protocol (PP) set 1 for TAVR care pathway for the Main Protocol and the attempted implant set for the FX Addendum.
  PP set 1 for TAVR care pathway consists of all implanted subjects with percutaneous and transfemoral access only and no concomitant procedures including percutaneous coronary intervention.
  Main Protocol and FX Addendum results are analyzed separately.
Measure: Median (Full Range); unit: Days
Arm/Group | Main Protocol | FX Addendum
Number analyzed (Participants) | 635 | 149
Days | 2.0 [1.0 to 31.0] | 1.0 [1.0 to 27.0]

3. Secondary Outcome: Aortic Regurgitation (AR)
Description: Percentage of subjects with ≥ moderate AR at discharge
Time Frame: Through discharge up to 7 days post index procedure.
Population: The implanted set was the basis for the AR secondary outcome measure for both the Main Protocol and FX Addendum.
  The implanted set consists of all the attempted implant subjects who are actually implanted with the Medtronic TAV device.
  Main Protocol and FX Addendum results are analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Protocol | FX Addendum
Number analyzed (Participants) | 627 | 145
Participants | 0 | 0

4. Secondary Outcome: Pacemaker Implantation or Worsening Conduction Disturbance
Description: Rate of pacemaker implant for new onset or worsening conduction disturbance at 30 days
Time Frame: 30 days
Population: The basis for the pacemaker implantation or worsening conduction disturbance secondary outcome measure was the PP set 2 for the Main Protocol and the attempted implant set for the FX Addendum.
  PP set 2 for conduction disturbance pathway set consists of all attempted implant subjects whose peri- and post-TAVR index procedure follows the conduction disturbance pathway management and cusp overlap technique.
  Main Protocol and FX Addendum results are analyzed separately.
Measure: Number; unit: Percent of Participants (K-M Rate)
Arm/Group | Main Protocol | FX Addendum
Number analyzed (Participants) | 322 | 151
Percent of Participants (K-M Rate) | 6.5 | 6.7

5. Secondary Outcome: Depth of Implant (Evolut FX Only)
Description: Percentage of subjects with a Non-Coronary Cusp (NCC) depth of implant between 1.0 and 5.0 mm (Evolut FX Addendum Only)
Time Frame: 30 days
Population: The FX Addendum implanted set was the basis for the depth of implant outcome measure.
  The implanted set consists of all attempted implant subjects who are actually implanted with the Medtronic Evolut™ FX device.
Measure: Count of Participants; unit: Participants
Arm/Group | FX Addendum
Number analyzed (Participants) | 136
Participants | 83

6. Secondary Outcome: Canting (Evolut FX Addendum Only)
Description: Percentage of subjects with a canting absolute value [NCC- Left Coronary Cusp(LCC)] of ≤ 2.0 mm (Evolut FX Addendum Only)
Time Frame: 30 Days
Population: The FX Addendum implanted set was the basis for the canting outcome measure.
  The implanted set consists of all attempted implant subjects who are actually implanted with the Medtronic Evolut™ FX device.
Measure: Count of Participants; unit: Participants
Arm/Group | FX Addendum
Number analyzed (Participants) | 135
Participants | 59

ADVERSE EVENTS:
Time Frame: Adverse Events collected starting at the time the informed consent was signed until the end of the study (i.e. 12 month follow-up post procedure) or study exit, whichever occurs first.
Description: Serious adverse events (SAE), device deficiencies (DD), and non-serious VARC-2 adverse events (that are outlined in the protocol) will be collected from the time of enrollment until the end of the study or until study exit, whichever comes first. Results reported below are through 12-month follow-up post procedure or study exit whichever occurs first.
  *Note there were no non-serious events by MedDRA preferred term that exceeded the 5% frequency threshold reporting.*
Arm/Group | Main Protocol | FX Addendum
All-Cause Mortality (participants affected / at risk) | 32/653 | 7/151
Serious Adverse Events (participants affected / at risk) | 212/653 | 44/151
Other Adverse Events (participants affected / at risk) | 0/653 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Protocol (N=653) | FX Addendum (N=151)
Anaemia (Blood and lymphatic system disorders) | 12 (15) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 3 (4)
Acute myocardial infarction (Cardiac disorders) | 17 (20) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 29 (34) | 7 (7)
Atrial flutter (Cardiac disorders) | 4 (4) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 55 (55) | 9 (10)
Atrioventricular block first degree (Cardiac disorders) | 6 (6) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 12 (12) | 1 (1)
Atrioventricular dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 3 (3)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 21 (21) | 4 (4)
Cardiac arrest (Cardiac disorders) | 9 (9) | 2 (2)
Cardiac failure (Cardiac disorders) | 8 (10) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 13 (14) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (6) | 3 (3)
Cardiac tamponade (Cardiac disorders) | 3 (3) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery embolism (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Defect conduction intraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Rhythm idioventricular (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 5 (5) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (8) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Device embolisation (General disorders) | 2 (2) | 1 (1)
Gravitational oedema (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Prosthetic cardiac valve regurgitation (General disorders) | 1 (1) | 0 (0)
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 0 (0)
Puncture site haemorrhage (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lung transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 12 (12) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cardiac valve vegetation (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (4) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Human anaplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (14) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Prosthetic valve endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic cerebral embolism (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 4 (4) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (9) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 10 (10) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 22 (22) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Electric shock sensation (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 4 (4) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 7 (7) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 4 (6)
Tongue paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 5 (5)
Device dislocation (Product Issues) | 4 (4) | 0 (0)
Device failure (Product Issues) | 2 (2) | 0 (0)
Lead dislodgement (Product Issues) | 1 (1) | 0 (0)
Prosthetic cardiac valve malfunction (Product Issues) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 9 (11) | 5 (5)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Disease risk factor (Social circumstances) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 2 (2) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Blue toe syndrome (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 1 (1)
Haemorrhage (Vascular disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 5 (6) | 3 (3)
Iliac artery dissection (Vascular disorders) | 3 (3) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Vascular dissection (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (8):
  • Study Protocol: Version 3.0 (2019-07-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_000.pdf
  • Study Protocol: Version 4.0 (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_001.pdf
  • Study Protocol: Version 5.0 (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_002.pdf
  • Study Protocol: Version 6.0 (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_003.pdf
  • Study Protocol: FX Addendum Version 1.0 (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_004.pdf
  • Study Protocol: FX Addendum Version 2.0 (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_005.pdf
  • Study Protocol: FX Addendum Version 3.0 (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/Prot_006.pdf
  • Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04091048/SAP_007.pdf